CLINICAL TRIAL: NCT01454440
Title: A RANDOMIZED TRIAL COMPARING EPTIFIBATIDE AND PLACEBO IN PATIENTS WITH DIFFUSE CORONARY DISEASE UNDERGOING DRUG-ELUTING STENTING
Brief Title: The INtegrilin Plus STenting to Avoid Myocardial Necrosis Trial (INSTANT)
Acronym: INSTANT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was stopped prematurely due to slow enrolment without code breaking.
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Giuseppe Biondi Zoccai, Assistant Professor in Cardiology, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2007-002617-39
Record Dates: First submitted 2011-10-06; First posted 2011-10-19 (Estimated); Last update posted 2011-10-19 (Estimated); Status verified 2011-10

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; Eptifibatide; Percutaneous coronary intervention; stable coronary artery disease; percutaneous coronary intervention (PCI); DES
MeSH Terms: conditions — Coronary Artery Disease | interventions — Eptifibatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Eptifibatide (Experimental): Intravenous eptifibatide (double bolus [180 microg/kg] followed by infusion [2 microg/kg per minute] for 18 to 24 hours after the procedure).
  Interventions: Drug: Eptifibatide
- Placebo (Placebo Comparator)
  Interventions: Drug: Eptifibatide

INTERVENTIONS:
Drug: Eptifibatide — Intravenous eptifibatide (double bolus [180 microg/kg] followed by infusion [2 microg/kg per minute] for 18 to 24 hours after the procedure) vs placebo.

SUMMARY:
Patients with stable coronary artery disease, undergoing PCI by means of implantation of >33 mm of DES, will be randomized single-blinded to eptifibatide plus unfractioned heparin according to the ESPRIT protocol vs placebo plus unfractioned heparin.

DETAILED DESCRIPTION:
BACKGROUND: Despite the availability of several potent antithrombotic agents, the optimal antiplatelet regimen in elective patients undergoing complex percutaneous coronary interventions is still debated. Aim of the INtegrilin plus STenting to Avoid myocardial Necrosis Trial (INSTANT) will be to assess the safety and efficacy of routine usage of the glycoprotein IIb/IIIa inhibitor eptifibatide in subjects already treated with aspirin and clopidogrel, and undergoing implantation of at least 2 drug-eluting stents in the same lesion, thus identifying a clinically stable but anatomically complex patient subset.

DESIGN: This will be a single-blind, placebo-controlled multicenter randomized trial METHODS: Patients with stable coronary artery disease, undergoing percutaneous coronary intervention (PCI) by means of implantation of >33 mm of DES (eg with two 23-mm DES, or one 32-mm and one 12-mm DES), will be randomized, after administration of aspirin and clopidogrel (600 mg loading dose recommended), to eptifibatide and unfractioned heparin according to the ESPRIT protocol vs placebo and unfractioned heparin. Blood draws for CK-MB mass, total CK and cardiac troponin levels will be taken at baseline, 6 and 12 hours post-procedurally. Patients will be followed for clinical events by direct visit or phone contact up to 6 months. The primary end-point of the study will be the rate of abnormal post-PCI CK-MB mass values. Secondary end-points will be: the composite of cardiac death, non-fatal myocardial infarction (MI), urgent target vessel revascularization (TVR), and thrombotic bailout GpIIb/IIIa inhibitor therapy within 180 days, and in-hospital, 1-month and 6-month major adverse cardiovascular events (MACE), defined as the composite of cardiac death, non-fatal MI, or urgent TVR.

IMPLICATIONS: The INSTANT Study will test for the first time the beneficial impact of routine GpIIb/IIIa inhibition on top of double oral antiplatelet treatment in clinically stable yet anatomically complex patients undergoing DES-implantation. Results of this single-blind randomized trial will provide important insights to improve the management strategy of patients and outcomes in the current DES era.

ELIGIBILITY:
Inclusion Criteria:

* male or female able to understand and sign a witnessed informed consent,
* age ≥ 18 years
* patients with stable (Canadian Cardiovascular Society I-IV) or unstable angina pectoris (but with the most recent anginal episode occurring >48 hours before the procedure [provided that the most recent CK-MB mass levels are within the limits of normal]) or documented silent ischemia
* stable hemodynamic conditions (systolic blood pressure>100, heart rate>40 and <100)
* no clinical and ECG changes suggestive of ongoing acute or recent (<48 hours) myocardial infarction.

Exclusion Criteria:

* female sex with childbearing potential
* age <18 years
* ongoing or recent episode (<48 hours) of unstable coronary artery disease (including both ST-elevation and non-ST-elevation acute coronary syndromes) without normalization of CK-MB mass levels
* administration of any GP IIb/IIIa inhibitors during the previous 2 weeks,
* serum creatinine >2.5 mg/dl or > 350 micromols/l
* ongoing serious bleeding or bleeding diathesis
* previous stroke in the last 6 months
* major surgery within the previous 6 weeks
* platelet count <100,000 per mm3
* ejection Fraction below 30%
* known hypersensitivity or contraindication to aspirin, heparin, clopidogrel or sensitivity to contrast which cannot be adequately pre-medicated
* hemodynamic instability (systolic blood pressure<100 mm Hg; heart rate<40 bpm or >100 bpm; complex ventricular arrhythmias; atrioventricular block) requiring balloon counterpulsation or inotropic support
* simultaneous participation in another device or drug study (patient must have completed the follow-up phase of any previous study at least 30 days prior to enrollment in this study)
* positive clinical history for intracranial neoplasia, arterio-venous malformation, aneurysm
* INR ≥ 2.0 or prothrombin time 1.2 times upper limit of normality
* clinically manifested reduced liver function
* programmed surgery within one month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2007-10; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Abnormal CK-MB level post-PCI | 2 weeks
  The primary end point will be the rate of elevated post-procedural peak CK-MB mass ratio values (ie above the upper limit of normal [ULN], eg 1.01*ULN, according to each participating hospital laboratory).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Turin, Turin, TO, Italy

REFERENCES:
- [Derived] Biondi-Zoccai G, Valgimigli M, Margheri M, Marzocchi A, Lettieri C, Stabile A, Petronio AS, Binetti G, Bolognese L, Bellone P, Sardella G, Contarini M, Sheiban I, Marra S, Piscione F, Romeo F, Colombo A, Sangiorgi G. Assessing the role of eptifibatide in patients with diffuse coronary disease undergoing drug-eluting stenting: the INtegrilin plus STenting to Avoid myocardial Necrosis Trial. Am Heart J. 2012 May;163(5):835.e1-7. doi: 10.1016/j.ahj.2012.02.009. PMID 22607870